CLINICAL TRIAL: NCT06959563
Title: Conducting an Early Phase Clinical Trial to Assess for HPV Antigen Presentation Therapeutic Biological Product Mix Activity That Suggests the Potential for Clinical Benefits of HPV Patients
Brief Title: Early Phase Clinical Trial About Therapeutic Biological Product Mix for Treating HPV
Acronym: 9vHPV-BCG
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair (Industry)
Collaborators: UnitedHealthcare (Other)
Responsible Party: Sponsor-Investigator, Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair, M.D., Ph.D., FAPCR, Sponsor-Investigator, Medical Director, IORG Director, Medical Monitor, Safety Officer, IRB Chair, Medicine Invention Design, Inc
Organization: Medicine Invention Design, Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IND 169135; IND 169135 (Registry Identifier: FDA, Investigational New Drug Application (IND)); NPI-1831468511 (Registry Identifier: HHS, Health Care Provider Individual); NPI-1023387701 (Registry Identifier: HHS, Health Care Provider Organization); FWA00015357 (Registry Identifier: HHS, Human Protections Administrator); IORG0007849 (Registry Identifier: HHS, IORG); IRB00009424 (Registry Identifier: HHS, IRB)
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: HPV Infection
Keywords: HPV; Antigen Presentation; APC; IGRA; Trained Immunity; Innate Immune Memory; Cervical
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
  * Single Usage
  * Single Dosage
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Assess for HPV Antigen Presentation (Experimental): Therapeutic Biological Product Mix activity 9vHPV Vaccine 1.0 mL add into BCG Organism 50 MG
  Interventions: Biological: 9vHPV Vaccine plus BCG Vaccine Mix for percutaneous use

INTERVENTIONS:
Biological: 9vHPV Vaccine plus BCG Vaccine Mix for percutaneous use — By the percutaneous route with the multiple puncture device - 9vHPV Vaccine 1.0 mL plus BCG Organism 50 MG Mix
  Other Names: 9vHPV Vaccine plus BCG Organism Mix

SUMMARY:
Conducting an early phase clinical trial to assess HPV Antigen Presentation Therapeutic Biological Product Mix activity that suggests the potential for clinical benefit of HPV patients.

1. Treat Infection of Multiple HPV Virus Strains via Trained Immunity.
2. Activate human HPV Antigen Presentation Reaction.
3. The human antigen presenting cells (APCs) can treat the HPV virus protein antigens into small peptide fragments, and then clear HPV virus in vivo.

DETAILED DESCRIPTION:
* Conducting an early phase clinical trial to assess HPV Antigen Presentation Therapeutic Biological Product Mix activity that suggests the potential for clinical benefit of HPV patients
* 20 Cervical HPV Infection Patients
* Positive testing HPV by standard PCR assay
* HPV infection without symptoms
* No clinical signs indicative of oncology
* TB negative participant is negative IGRA blood test with TB antigens
* 9vHPV Vaccine 1.0 mL plus BCG Organism 50 MG Mix
* By the percutaneous route with the multiple puncture device
* Negative testing HPV by standard PCR assay after percutaneous 21 days
* Positive IGRA blood test with HPV protein antigen after percutaneous use 21 days
* Our trial duration will be 12-week duration.

ELIGIBILITY:
Conducting an early phase clinical trial to assess HPV Antigen Presentation Therapeutic Biological Product Mix that suggests the potential for clinical benefit of HPV patients.

20 Cervical HPV Infection Patients

Inclusion Criteria:

* Cervical HPV Infection Patients
* Positive testing HPV by standard PCR assay
* HPV infection without symptoms
* No clinical signs indicative of oncology
* TB negative participant is negative IGRA blood test with TB antigens

Exclusion Criteria:

* Pregnant
* Thrombosis
* Bleeding
* Allergy
* TB positive participant is positive IGRA blood test with TB antigens
* Symptoms of HPV infection
* Clinical signs suggestive of other infection
* Symptoms suggestive of other infection
* Clinical signs indicative of oncology
* Evidence of critical illness

Ages: 24 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Cervical is a female organ.
Enrollment: 20 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2026-09-18 (Estimated); Study Completion 2026-09-28 (Estimated)

PRIMARY OUTCOMES:
20 HPV Participants with HPV testing by standard PCR assay | Duration at least 28 days
  Negative testing HPV by standard PCR assay after percutaneous 21 days
20 HPV Participants with IGRA blood test with HPV protein antigen | Duration at least 28 days
  Positive IGRA blood test with HPV protein antigen after percutaneous use 21 days
20 HPV Participants with IGRA blood test with TB antigens | Duration at least 28 days
  * Negative IGRA blood test with TB antigens before percutaneous use
  * Positive IGRA blood test with TB antigens after percutaneous use 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Han ID Xu, MD/PhD/FAPCR, Study Chair — Medicine Invention Design Incorporation; Han Xu, MD/PhD/FAPCR, Study Director — Medicine Invention Design Incorporation; Han Xu, MD/PhD/FAPCR, Principal Investigator — Medicine Invention Design Incorporation
Locations (1):
- Medicine Invention Design, Inc., Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: IORG0007849 — http://ohrp.cit.nih.gov/search/search.aspx?styp=bsc
- See also: IRB00009424 — http://ohrp.cit.nih.gov/search/search.aspx?styp=bsc
- See also: FWA00015357 — http://ohrp.cit.nih.gov/search/search.aspx?styp=bsc

DOCUMENTS (3):
  • Study Protocol (2025-05-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT06959563/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT06959563/SAP_001.pdf
  • Informed Consent Form (2025-05-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT06959563/ICF_002.pdf